CLINICAL TRIAL: NCT07200687
Title: Effects of Combined Music Therapy and Occupational Therapy on Motor and Physiological Parameters in Children With Neurological Impairments: A Non-Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armakola Filomeni (Other)
Responsible Party: Sponsor-Investigator, Armakola Filomeni, MD, MSc, PhDc, University of West Attica
Organization: University of West Attica (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA.D.A.-AR.PROT: 66741
Record Dates: First submitted 2025-09-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Palsy (CP); Encephalitis; Brain Tumor (After Recovery)
MeSH Terms: conditions — Cerebral Palsy; Encephalitis; Brain Neoplasms | interventions — Music Therapy; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Occupational Therapy + Music Therapy (with scoliosis) (Experimental): This arm includes children with neurological conditions and scoliosis who will receive a structured occupational therapy program incorporating music therapy elements
  Interventions: Other: Music therapy; Other: occupational therapy
- Occupational Therapy (Active Comparator): This group includes children with similar neurological conditions and scoliosis who will receive the same occupational therapy program without any music therapy integration.
  Interventions: Other: occupational therapy
- Occupational Therapy + Music Therapy (no scoliosis) (Experimental): Children with neurological conditions but without scoliosis receive the same occupational therapy program combined with music therapy. This arm allows the evaluation of music therapy's effects in children with neurological conditions independent of spinal deformity
  Interventions: Other: Music therapy; Other: occupational therapy

INTERVENTIONS:
Other: Music therapy — this research hopes to offer new insights into the benefits of combining music therapy with occupational therapy.
  Arms: Occupational Therapy + Music Therapy (no scoliosis); Occupational Therapy + Music Therapy (with scoliosis)
Other: occupational therapy — standard treatment

SUMMARY:
This study aims to explore the effects of an occupational therapy program combined with music therapy elements on children 5-12 years old with neurological disorders including those with neurogenic scoliosis. Occupational therapy programs typically focus on improving motor and cognitive functions to enhance the child's overall participation and daily functioning. Music has been shown to positively affect brain areas involved in emotions, memory, and language, and may reduce stress and increase feelings of happiness.

The study will measure changes in biological markers such as blood pressure, oxygen saturation, heart rate, and respiratory rate, as well as improvements in functionality for upper limbs but also balance and walking ability after the therapy program. These markers can provide valuable information about the physical health and quality of life of the children, which is currently lacking for the Greek population.

By investigating these biological indicators along with functional outcomes, this research hopes to offer new insights into the benefits of combining music therapy with occupational therapy. This may encourage better engagement from families and support rehabilitation specialists in demonstrating the value of their interventions even before functional improvements become noticeable

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of a neurological condition with established neurological signs (e.g., motor or cognitive impairments)

* Cerebral Palsy (GMFCS levels I-II),
* Brain infections (e.g., encephalitis),
* Brain neoplasms
* Ability to follow simple instructions and participate in an occupational therapy program,
* Medical clearance to participate in physical activity

Exclusion Criteria:

* Degenerative neurological diseases,
* Metabolic disorders affecting the nervous system,
* Neuromuscular disorders, including muscular dystrophy and congenital myopathies,
* Peripheral nervous system damage,
* Current use of corticosteroids,
* Botulinum toxin injection within 30 days prior to the intervention program,
* Hearing loss or diagnosed deafness

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
10M WALK TEST | From enrollment to the end of treatment at 6weeks
  WALKING ABILITY
pediatric balance scale | "From enrollment to the end of treatment at 6 weeks"
  balance Pediatric Balance Scale (PBS) is used, specifically the Greek validated version ("Pediatric Balance Scale - Greek version," PBS-GR), as translated and cross-culturally adapted by Bania et al. (2023). The scale ranges from 0 to 56, with higher scores indicating better balance performance and a better outcome. The PBS-GR has been shown to have high interrater reliability in children with movement impairment

SECONDARY OUTCOMES:
blood pressure | Arterial blood pressure will be measured using an automated electronic sphygmomanometer (mmHg). Measurements will be taken in a seated position after 5 minutes of rest, immediately before and immediately after (45 min) each therapy session.
  PHYSIOLOGICAL BIOMARKERS
SaO2 oxygen saturation | Oxygen saturation will be measured non-invasively using a fingertip pulse oximeter (%). Measurements will be taken in a seated position, after 5 minutes of rest, immediately before and immediately after each (45 min) therapy session.
  physiological marker
heart rate | Heart rate will be measured non-invasively using an electronic sphygmomanometer (beats per minute, bpm). Measurements will be taken in a seated position, after 5 minutes of rest, immediately before and immediately after (45 min)each therapy session
  physiological marker
Respiratory Rate | Respiratory rate will be measured manually by counting visible thoracic movements (breaths per minute) for 60 seconds while the child is in a seated position before and after (45 min) each therapy session
  physiological marker

CONTACTS AND LOCATIONS:
Locations (1):
- Athens Children's Hospital P.&A. Kiriakou, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No